CLINICAL TRIAL: NCT03490292
Title: Phase I/II Trial of Avelumab in Combination With Chemoradiation in the Treatment of Stage II/III Resectable Esophageal and Gastroesophageal Cancer
Brief Title: Avelumab With Chemoradiation for Stage II/III Resectable Esophageal and Gastroesophageal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW17106; NCI-2018-00150 (Registry Identifier: NCI Trial ID); 2017-1491 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 7/5/2021 (Other: UW Madison)
Record Dates: First submitted 2018-02-09; First posted 2018-04-06 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Resectable Esophageal Cancer; GastroEsophageal Cancer
MeSH Terms: interventions — Chemoradiotherapy; Carboplatin; Paclitaxel; Radiation

STUDY DESIGN:
Intervention Model Description: The study is a two-part phase 1/2 clinical trial conducted in one center.
  Part 1. Run-in phase to assess the safety and tolerability of avelumab in combination with chemoradiation. Will enroll 6 patients, after which accrual will be stopped temporarily while safety data is being obtained.
  Part 2. An open-label phase 2 study. Part 2 will obtain further safety data of the proposed drug combination and will evaluate the anti-tumor efficacy of perioperative avelumab and chemoradiation in this patient population. Will enroll 18 additional patients.
  Each phase of the study will have a 21-day screening period, treatment procedures (neoadjuvant therapy, resection and adjuvant therapy), and active surveillance for a year after the completion of adjuvant therapy.
  After active surveillance visit at 12 months post treatment completion, survival data and disease status will be collected via phone calls or medical record review every 6 months during the following 3 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Run-In Phase (Experimental): 6 patients enrolled will receive weekly carboplatin (AUC2) and paclitaxel (50 mg/m2) [intravenous infusion on days 1, 8, 15, 22, & 29] while undergoing radiation therapy [23 fractions, M-F, estimated completion day 35].
  Avelumab combined with Chemoradiation - Avelumab (10 mg/kg IV) every 2 weeks starting on the day of the last chemotherapy infusion (day 29). A total of 3 doses administered during the pre-operative period and an additional 6 doses of avelumab post-operatively.
  Trial enrollment will resume after at least 5 patients do not have a dose-limiting toxicity (DLT) during the DLT evaluation period or until all 6 patients are seen for post-operative evaluation. If 2 or more patients experience dose limiting toxicities associated with the proposed treatments, further accrual of the subjects will be halted and trial will be suspended. Trial may be reopened in the future with appropriate schedule and dose modifications of the proposed treatment.
  Interventions: Combination Product: Avelumab combined with Chemoradiation; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation
- Expansion Cohort (Experimental): Following a determination of safe and tolerable treatment outcome of the Run-In Phase, Part 2 of the trial will enroll 18 additional patients to evaluate activity of the proposed treatment and to obtain further safety information (carboplatin, paclitaxel, radiation & Avelumab combined with Chemoradiation).
  Interventions: Combination Product: Avelumab combined with Chemoradiation; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation

INTERVENTIONS:
Combination Product: Avelumab combined with Chemoradiation — Co-administration of avelumab with chemoradiation in pre-operative period.
Drug: Carboplatin — Weekly Carboplatin (AUC2) [intravenous infusion on days 1, 8, 15, 22, & 29]
Drug: Paclitaxel — Weekly paclitaxel [intravenous infusion on days 1, 8, 15, 22, & 29]
Radiation: Radiation — Radiation therapy [23 fractions, M-F, estimated completion day 35]

SUMMARY:
This is a 2 part Phase I/II clinical trial evaluating the safety, tolerability and efficacy of avelumab in combination with chemoradiation in patients with resectable esophageal and gastroesophageal cancer.

Part 1: This is the run-in phase of the trial. This portion will determine the safety and tolerability of avelumab in combination with chemoradiotherapy in 6 patients. The proposed combination will be considered as safe if dose limiting toxicities are observed in at most 1 patient.

Part 2: This is a Phase 2 portion of the trial, which will evaluate the efficacy of the proposed treatment regimen in patients with stage II/III resectable esophageal and gastroesophageal cancer

DETAILED DESCRIPTION:
Background:

Neoadjuvant chemoradiation is part of the standard of care for patients with stage II and III resectable esophageal and gastroesophageal cancer. This approach is based on the results of a large randomized clinical trial (CROSS) that demonstrated superior survival in patients receiving neoadjuvant chemoradiotherapy followed by surgical resection compared to patients treated with surgery alone. Pathological complete response at the time of resection is strongly linked to better survival. However, with current strategies pathological complete response is achieved only in a minority (29%) of patients. Remaining patients, especially those with positive lymph nodes at the time of the resection, are at significant risk for recurrences. Five-year survival rate for these patients is only 37%, and overall survival is as low as 9 months for those with persistent lymph node disease. Among patients who develop recurrent disease, most present with distant metastases outside of the radiation field. This is not surprising since the accepted treatment paradigm for this disease does not target possible disseminated microscopic systemic disease. Hence, novel strategies are needed to improve outcomes of these patients. We propose conducting a phase I/II clinical trial evaluating a role of immune checkpoint inhibitor in combination with chemoradiotherapy and post-operatively in the management of resectable esophageal cancer.

Study Rationale:

1. A number of preclinical and clinical studies demonstrated synergism between radiation and immunotherapy, suggesting that combining these approaches can enhance anti-tumor activity and increase treatment efficacy.
2. Immune checkpoint inhibitors have demonstrated promising activity in a subset of patients with metastatic esophageal and gastric cancers. Moving these agents into neoadjuvant setting may increase the cure rate of this disease compared to the standard approach.
3. Current neoadjuvant therapy does not target any potential microscopic disease outside of the radiation field since chemotherapy serves primarily as a radiation sensitizer. Immunotherapy treatment will target both local and systemic disease.

Hypothesis:

We hypothesize that co-administration of avelumab with chemoradiation will be well tolerated and will increase pathological complete response rate in resected tumor specimens. We hypothesize that avelumab treatment will also decrease the rates of disease recurrence.

Study Design:

This is a 2 part Phase I/II clinical trial evaluating the safety, tolerability and efficacy of avelumab in combination with chemoradiation in patients with resectable esophageal and gastroesophageal cancer.

Part 1: This is the run-in phase of the trial. This portion will determine the safety and tolerability of avelumab in combination with chemoradiotherapy in 6 patients. The proposed combination will be considered as safe if dose limiting toxicities are observed in at most 1 patient.

Part 2: This is a Phase 2 portion of the trial, which will evaluate the efficacy of the proposed treatment regimen in patients with stage II/III resectable esophageal and gastroesophageal cancer.

Objectives:

Primary: Evaluate the safety of avelumab in combination with chemoradiation in patients with resectable esophageal cancer and gastroesophageal receiving perioperative therapy.

Secondary: Obtain efficacy data and further safety data of the proposed drug combination in this patient population.

Exploratory objectives: The translational focus of the study will evaluate changes in tumor microenvironment that occur in response to radiation and immunotherapy.

Endpoints:

Part 1 - Primary endpoint: Establish safety and tolerability of the proposed treatment.

Part 2 - Primary Endpoint: Pathological complete response rate.

Part 2 - Secondary Endpoints:

1. Safety and tolerability.
2. Disease free survival.
3. Incidence of surgical complications.
4. Rate of R0 resection.

Number of centers & patients: One center.

Part 1: total of 6 eligible patients will be accrued to evaluate the safety and tolerability of the proposed combination.

Part 2: 18 patients will be enrolled in the phase 2 portion of the trial.

Population:

Patients with histologically confirmed, potentially curable squamous-cell carcinoma, adenocarcinoma, or large-cell undifferentiated carcinoma of the esophagus and gastroesophagus who are candidates for neoadjuvant therapy and surgical resection.

Investigational drugs:

Avelumab (Provided by EMD Serono). IND information to be added as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed, potentially curable squamous-cell carcinoma, adenocarcinoma, or large-cell undifferentiated carcinoma of the esophagus and gastroesophagus (Siewert type 1-3)
2. Locoregional disease with clinical stage of T1N1 or T2-3N0-2
3. No clinical evidence of metastatic spread. Staging should include endoscopic ultrasound and positron emission tomography/computed tomography (PET/CT) as recommended by National Comprehensive Cancer Network (NCCN) guidelines. PET/CT should be performed within 3 weeks of signing informed consent
4. Age 18 years or older
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Subjects must be deemed to be potential surgical candidates by an evaluating surgeon
7. Adequate organ function:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Hemoglobin ≥ 9 g/dL (transfusions allowed)
   3. Platelets ≥ 100 x 109/L
   4. Aspartate transaminase/Alanine transaminase (AST/ALT) ≤ 2.5 x ULN
   5. Total serum bilirubin of ≤1.5 x institutional upper limit of normal (ULN)
   6. Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula
8. Female patients of childbearing potential must have a negative pregnancy test (urine or serum) within 21 days prior to the start of the study drug treatment and must agree to use adequate birth control if conception is possible during the study and up to 30 days after the completion of adjuvant therapy
9. Male patients must agree to use adequate birth control during the study and up to 30 days after the last avelumab dose
10. Women who are nursing must discontinue breast-feeding prior to the enrollment in the trial
11. Patient must be able and willing to comply with study procedures as per protocol
12. Patient able to understand and willing to sign and date the written voluntary informed consent form (ICF) at screening visit prior to any protocol-specific procedures

Exclusion Criteria:

1. Prior history of radiation to the mediastinum
2. Diagnosis of cervical esophageal carcinoma
3. Other active malignancy within the last 3 years (except for non-melanoma skin cancer, a non-invasive/in situ cancer, or indolent non metastatic Gleason 6 prostate cancer)
4. Subjects with an active or known autoimmune disease. Subjects with type I diabetes mellitus, hypo- or hyperthyroidism only requiring hormone replacement/suppression, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic immunosuppressive treatment are eligible
5. Current use of immunosuppressive medication, except for the following:

   1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
   2. systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent
   3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
6. Active infection requiring systemic therapy at the time of study treatment initiation
7. Prior organ transplantation including allogenic stem-cell transplantation
8. Known history of testing positive for HIV or known immunodeficiency syndrome
9. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
10. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines
11. Major surgery within prior 4 weeks of treatment initiation (the surgical incision should be fully healed prior to all neoadjuvant treatment initiation)
12. Any prior anticancer therapy for esophageal cancer
13. History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin, paclitaxel or avelumab, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3)
14. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication. Patients with stable rate-controlled atrial fibrillation will be allowed to participate
15. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
16. Psychological, familial, or sociological condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Uboha, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Wisconsin Hospital and Clinics from May 2018 through June 2021.
Groups:
- Run In Phase: 6 patients enrolled will receive weekly carboplatin (AUC2) and paclitaxel (50 mg/m2) [intravenous infusion on days 1, 8, 15, 22, & 29] while undergoing radiation therapy [23 fractions, M-F, estimated completion day 35].
  Avelumab combined with Chemoradiation - Avelumab (10 mg/kg IV) every 2 weeks starting on the day of the last chemotherapy infusion (day 29). A total of 3 doses administered during the pre-operative period and an additional 6 doses of avelumab post-operatively.
  Trial enrollment will resume after at least 5 patients do not have a dose-limiting toxicity (DLT) during the DLT evaluation period or until all 6 patients are seen for post-operative evaluation. If 2 or more patients experience dose limiting toxicities associated with the proposed treatments, further accrual of the subjects will be halted and trial will be suspended. Trial may be reopened in the future with appropriate schedule and dose modifications of the proposed treatment.
  Avelumab combined with Chemoradiation: Co-administration of avelumab with chemoradiation in pre-operative period.
  Carboplatin: Weekly Carboplatin (AUC2) [intravenous infusion on days 1, 8, 15, 22, & 29]
  Paclitaxel: Weekly paclitaxel [intravenous infusion on days 1, 8, 15, 22, & 29]
  Radiation: Radiation therapy [23 fractions, M-F, estimated completion day 35]
- Expansion Cohort: Following a determination of safe and tolerable treatment outcome of the Run-In Phase, Part 2 of the trial will enroll up to 18 additional patients to evaluate activity of the proposed treatment and to obtain further safety information (carboplatin, paclitaxel, radiation & Avelumab combined with Chemoradiation).
  Avelumab combined with Chemoradiation: Co-administration of avelumab with chemoradiation in pre-operative period.
  Carboplatin: Weekly Carboplatin (AUC2) [intravenous infusion on days 1, 8, 15, 22, & 29]
  Paclitaxel: Weekly paclitaxel [intravenous infusion on days 1, 8, 15, 22, & 29]
  Radiation: Radiation therapy [23 fractions, M-F, estimated completion day 35]
Period: Treatment: Run-In Phase (June-Oct 2018)
Arm/Group | Run In Phase | Expansion Cohort
Started | 6 | 0
Completed | 6 | 0
Not Completed | 0 | 0
Period: Interim Analysis
Arm/Group | Run In Phase | Expansion Cohort
Started (Run-In Phase Participants analyzed for Dose Limiting Toxicities) | 6 | 0
Completed | 6 | 0
Not Completed | 0 | 0
Period: Treatment: Expansion (Feb 2019-Dec 2021)
Arm/Group | Run In Phase | Expansion Cohort
Started | 0 | 16
Completed | 0 | 9
Not Completed | 0 | 7
Not completed — Death | 0 | 1
Not completed — Off Treatment Pre-Surgery | 0 | 2
Not completed — Off Treatment Post-Surgery | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: 1 Year Follow Up Post Last Dose
Arm/Group | Run In Phase | Expansion Cohort
Started | 6 | 9
Completed | 5 | 8
Not Completed | 1 | 1
Not completed — Death | 1 | 1
Period: Survival Follow up 4 Yr Post Last Dose
Arm/Group | Run In Phase | Expansion Cohort
Started | 5 | 8
Completed | 5 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Run-In Phase: 6 patients enrolled will receive weekly carboplatin (AUC2) and paclitaxel (50 mg/m2) [intravenous infusion on days 1, 8, 15, 22, & 29] while undergoing radiation therapy [23 fractions, M-F, estimated completion day 35].
- Expansion Cohort: Following a determination of safe and tolerable treatment outcome of the Run-In Phase, Part 2 of the trial will enroll up to 18 additional patients to evaluate activity of the proposed treatment and to obtain further safety information (carboplatin, paclitaxel, radiation & Avelumab combined with Chemoradiation).
- Total: Total of all reporting groups
Arm/Group | Run-In Phase | Expansion Cohort | Total
Number analyzed (Participants) | 6 | 16 | 22
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 0 | 2 | 2
  50-59 years | 2 | 2 | 4
  60-69 years | 3 | 5 | 8
  70-79 years | 1 | 7 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 6 | 14 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 15 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 16 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 16 | 22
Tumor Location [Count of Participants; unit: Participants]
  Esophageal | 0 | 8 | 8
  Gastroesophageal Junction | 6 | 8 | 14
Histology [Count of Participants; unit: Participants]
  Squamous | 0 | 3 | 3
  Adenocarcinoma | 6 | 13 | 19
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG)
  Participants
    0 - Fully active, able to carry on all pre-disease performance without restriction | 4 | 8 | 12
    1 - Restricted in strenuous activity, ambulatory, able to carry out light or sedentary work | 2 | 8 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity
Description: A total number of 6 subjects will be enrolled during the run-in phase of the trial. A sample size of 6 is sufficient to estimate the true dose limiting toxicity rate of the proposed avelumab/chemoradiation therapy with adequate accuracy.The proposed treatment combination will be considered as safe if dose limiting toxicities are observed in at most 1 patient.
Time Frame: Up to 4 weeks post-resection (up to approximately 4 months on study) of all Run-In Phase participants
Measure: Count of Participants; unit: Participants
Groups:
- Run-In Phase: 6 patients enrolled will receive weekly carboplatin (AUC2) and paclitaxel (50 mg/m2) [intravenous infusion on days 1, 8, 15, 22, & 29] while undergoing radiation therapy [23 fractions, M-F, estimated completion day 35].
  Avelumab combined with Chemoradiation - Avelumab (10 mg/kg IV) every 2 weeks starting on the day of the last chemotherapy infusion (day 29). A total of 3 doses administered during the pre-operative period and an additional 6 doses of avelumab post-operatively.
  Trial enrollment will resume after at least 5 patients do not have a DLT during the DLT evaluation period or until all 6 patients are seen for post-operative evaluation. If 2 or more patients experience dose limiting toxicities associated with the proposed treatments, further accrual of the subjects will be halted and trial will be suspended. Trial may be reopened in the future with appropriate schedule and dose modifications of the proposed treatment.
  Avelumab combined with Chemoradiation: Co-administration of avelumab with chemoradiation in pre-operative period.
  Carboplatin: Weekly Carboplatin (AUC2) [intravenous infusion on days 1, 8, 15, 22, & 29]
  Paclitaxel: Weekly paclitaxel [intravenous infusion on days 1, 8, 15, 22, & 29]
  Radiation: Radiation therapy [23 fractions, M-F, estimated completion day 35]
Arm/Group | Run-In Phase
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Number of Participants With Pathological Complete Response
Description: Pathologic compete response (pCR) is defined as an absence of any viable tumor at microscopic examination of the primary tumor and any lymph nodes sampled after surgery following neoadjuvant therapy. Participants with invalid/missing pCR assessments will be defined as non-responders. The number and frequency of patients with a pCR will be summarized in tabular format.
Time Frame: Post-resection (80-100 days) pathology review for all participants (up to approximately 4 months on study)
Population: 3 participants did not have surgery.
Measure: Count of Participants; unit: Participants
Groups:
- Run In Phase: Run-In Phase was to determine safe and tolerable treatment outcome (carboplatin, paclitaxel, radiation & Avelumab combined with Chemoradiation).
Arm/Group | Run In Phase | Expansion Cohort
Number analyzed (Participants) | 6 | 16
Participants | 2 | 3

3. Secondary Outcome: Number of Participants With Treatment Related Adverse Events Greater Than or Equal to Grade 3
Description: Part 2 will further evaluate the safety of the studied drug combination, building on the observations from Part 1.
  All patients who receive at least one dose of avelumab will be evaluated for toxicity. Toxicities observed will be summarized in terms of types and severities by Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 (see Adverse Events section).
Time Frame: Up to 30 days post-avelumab of all (up to 4 months on study)
Measure: Count of Participants; unit: Participants
Arm/Group | Run In Phase | Expansion Cohort
Number analyzed (Participants) | 6 | 16
Participants
  Lymphopenia | 5 | 16
  White Blood Cell Decrease | 4 | 9
  Neutropenia | 2 | 4
  Diarrhea | 0 | 1
  Acute Kidney Injury | 0 | 1
  Hypotension | 0 | 1
  Dehydration | 1 | 0
  Infusion Reaction | 0 | 1
  Nausea | 1 | 0
  Hypersensitivity Reaction to Avelumab | 0 | 1

4. Secondary Outcome: Number of Participants Who Did or Did Not Complete Planned Treatment
Description: Part 2 will further evaluate the tolerability of the studied drug combination, building on the observations from Part 1.
  Tolerability will be reported as the number of subjects who did or did not complete the planned treatment, including the reason they ended treatment early.
Time Frame: Up to 30 days post-avelumab of all participants (up to 4 months on study)
Measure: Count of Participants; unit: Participants
Groups:
- Run In Phase: Run-In Phase was to determine a safe and tolerable treatment outcome (carboplatin, paclitaxel, radiation & Avelumab combined with Chemoradiation).
Arm/Group | Run In Phase | Expansion Cohort
Number analyzed (Participants) | 6 | 16
Participants
  Completed All Protocol Treatment | 6 | 13
  Completed Neoadjuvant Therapy and Planned Surgical Resection | 6 | 10
  Did not complete all planned Neoadjuvant Treatment | 0 | 3

5. Secondary Outcome: Number of Participants With Unexpected Surgical Complications
Time Frame: Following resection (80 -100 days) for all participants (up to approximately 5 months on study)
Population: 3 participants did not undergo resection
Measure: Count of Participants; unit: Participants
Arm/Group | Run In Phase | Expansion Cohort
Number analyzed (Participants) | 6 | 13
Participants | 0 | 0

6. Secondary Outcome: Rate of R0 Resection
Description: R0 resection corresponds to resection for cure or complete remission.
Time Frame: Following pathology review post-resection (80 -100 days) for all participants (up to approximately 4 months on study)
Population: 3 participants did not have surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Run In Phase | Expansion Cohort
Number analyzed (Participants) | 6 | 13
Participants | 5 | 10

7. Secondary Outcome: Disease Free Survival
Description: Disease free survival (DFS) will be defined as the number of days from the day of resection to the day a subject experiences an event of disease recurrence or death, whichever comes first. If a subject has not experienced an event of disease recurrence progression or death at the time of analysis, then the subject's data will be censored at the date of the last available evaluation. DFS will be summarized using point estimates of the median time to progression and the associated 95% confidence interval. The data will be presented graphically using Kaplan-Meier plots.
Time Frame: Up to 4 years post-resection for all participants
Population: median disease free survival was not reached by data cut-off on 7/13/2023, 1-year estimated Kaplan-Meier RFS was determined and reported in a separate outcome measure, all participants received the same intervention and are reported as a single group
Measure: Median (Full Range); unit: days
Groups:
- Carboplatin, Paclitaxel, Radiation & Avelumab Combined With Chemoradiation: All participants had 21-day screening period, treatment procedures (neoadjuvant therapy, resection and adjuvant therapy), and active surveillance for a year after the completion of adjuvant therapy.
  After active surveillance visit at 12 months post treatment completion, survival data and disease status will be collected via phone calls or medical record review every 6 months during the following 3 years.
Arm/Group | Carboplatin, Paclitaxel, Radiation & Avelumab Combined With Chemoradiation
Number analyzed (Participants) | 22
days | NA [NA to NA] — median disease free survival was not reached by data cut-off on 7/13/2023, 1-year estimated Kaplan-Meier RFS was determined

8. Secondary Outcome: Estimated 1-year Recurrence Free Survival
Time Frame: up to 1 year
Population: 17 participants were evaluable for response assessment, all participants received the same intervention and are reported as a single group
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin, Paclitaxel, Radiation & Avelumab Combined With Chemoradiation
Number analyzed (Participants) | 17
percentage of participants | 71 [43 to 87]

ADVERSE EVENTS:
Time Frame: up to 4 weeks post resection (up to 4 months on study), survival data collected up to 4 years
Description: Participants in the Run-In Phase and the Expansion Cohort received the same treatment.
Groups:
- Run In Phase: Determination of safe and tolerable treatment outcome (carboplatin, paclitaxel, radiation & Avelumab combined with Chemoradiation).
- Expansion Cohort: Additional patients to evaluate activity of the proposed treatment and to obtain further safety information (carboplatin, paclitaxel, radiation & Avelumab combined with Chemoradiation).
Arm/Group | Run In Phase | Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 1/6 | 6/16
Serious Adverse Events (participants affected / at risk) | 3/6 | 10/16
Other Adverse Events (participants affected / at risk) | 6/6 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run In Phase (N=6) | Expansion Cohort (N=16)
Esophageal leak (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 2 (3)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Accidental J-tube removal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Colonic Ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run In Phase (N=6) | Expansion Cohort (N=16)
Esophagitis (Gastrointestinal disorders) | 3 (4) | 11 (13)
Constipation (Gastrointestinal disorders) | 4 (6) | 8 (13)
Nausea (Gastrointestinal disorders) | 3 (5) | 9 (18)
Diarrhea (Gastrointestinal disorders) | 3 (8) | 9 (18)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (12)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 5 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (33) | 15 (83)
White blood cell decreased (Investigations) | 6 (18) | 15 (57)
Neutrophil count decreased (Investigations) | 4 (9) | 12 (29)
Platelet count decreased (Investigations) | 5 (6) | 12 (19)
Weight loss (Investigations) | 4 (7) | 10 (24)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 4 (4)
Blood bicarbonate decreased (Investigations) | 0 (0) | 4 (6)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (5)
Creatinine increased (Investigations) | 0 (0) | 2 (5)
Thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 12 (22)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6) | 12 (29)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4) | 12 (22)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 6 (7)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (4) | 4 (11)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 14 (19)
Fever (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Generalized edema (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (8) | 11 (26)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 4 (5)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2)
Akathisia (Nervous system disorders) | 0 (0) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (5) | 7 (13)
Hypotension (Vascular disorders) | 1 (2) | 5 (7)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 6 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — accidental chest tube removal
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) — Sinus Infection
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 7 (9)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Head laceration
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Foot drop
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0) — thyroiditis
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Hepatocellular Carcinoma
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Perforated eardrum - left
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT03490292/Prot_SAP_000.pdf